CLINICAL TRIAL: NCT00511667
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Sequential Panel Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK0941 After Multiple Daily Administration of MK0941 Before Each Meal (q.a.c.) in Subjects With Type 2 Diabetes
Brief Title: A Multiple Dose Investigational Drug Study in Patients With Type 2 Diabetes (MK-0941-005)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0941-005; 2007_595
Record Dates: First submitted 2007-08-02; First posted 2007-08-06 (Estimated); Results first posted 2012-06-26 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 3-((6-(ethylsulfonyl)-3-pyridinyl)oxy)-5-(2-hydroxy-1-methylethoxy)-N-(1-methyl-1H-pyrazol-3-yl)benzamide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- MK0941 (Experimental)
  Interventions: Drug: MK0941
- Placebo (Placebo Comparator)
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: MK0941 — MK0941 10 mg, 20 mg, 30 mg, or 40 mg before each meal or before 2 meals each day, or 60 mg before 2 meals each day
  Arms: MK0941
Drug: Comparator: Placebo — Placebo 10 mg, 20 mg, 30 mg, or 40 mg before each meal or before 2 meals each day, or 60 mg before 2 meals each day
  Arms: Placebo

SUMMARY:
A multiple dose study to assess the safety and pharmacokinetics of an investigational drug in patients with type 2 diabetes. The primary hypotheses of the study are that multiple daily MK-0941 in subjects with T2DM with or without adequate control on metformin will be sufficiently safe and well tolerated to permit continued clinical investigation.

ELIGIBILITY:
Inclusion Criteria:

* Nonsmoking Male or Female (of non-child bearing potential)
* Diagnosis of Type 2 Diabetes and is being treated with diet and exercise alone or with less than 3 oral anti-hyperglycemic agents
* Panel E only (MK0941 60 mg before 2 meals each day): diagnosis of Type 2 Diabetes and is on a dose of metformin of greater than or equal to 1500 mg for 8 weeks or more

Exclusion Criteria:

* Subject is on insulin or a peroxisome proliferator-activated receptor (PPAR) agonist
* Subject is on 3 or more oral anti-diabetes medications
* Subject has a history of type 1 diabetes
* Subject has a diagnosis of glaucoma or is blind
* Subject has had trauma to one or both eyes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-0941: All participants receiving any dose of MK-0941
- Placebo: All participants receiving any dose of placebo
Period: Overall Study
Arm/Group | MK-0941 | Placebo
Started | 52 | 18
Completed | 40 | 15
Not Completed | 12 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Site terminated | 6 | 1
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-0941 | Placebo | Total
Number analyzed (Participants) | 52 | 18 | 70
Age, Customized [Number; unit: participants]
  29 to 70 years | 52 | 18 | 70
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 10 | 33
  Male | 29 | 8 | 37

OUTCOME MEASURES:

1. Primary Outcome: Participants With Any Clinical Adverse Experience
Time Frame: Approximately 30 days after last dose of study drug (14 days for participants receiving MK0941 40 mg before each meal)
Measure: Number; unit: percentage of of participants
Arm/Group | MK-0941 | Placebo
Number analyzed (Participants) | 52 | 18
percentage of of participants | 51.9 | 61.1

2. Secondary Outcome: Area Under the Concentration-time Curve (AUC0-24) of MK-0941 After Multiple Doses of MK0941
Time Frame: Up to 72 hours after dosing (up to 24 hours for participants receiving MK0941 60 mg before 2 meals each day)
Measure: Mean (Standard Deviation); unit: nM-hr
Groups:
- Panel A: MK-0941 10 mg: MK-0941 10 mg before each meal for 5 days. Sampling began after dosing on Day 5.
- Panel B: MK-0941 20 mg: MK-0941 20 mg before each meal for 5 days. Sampling began after dosing on Day 5.
- Panel C: MK-0941 40 mg Day 7: MK-0941 40 mg before each meal for 7 days. Sampling began after dosing on Day 7. These participants are different from those in Panel D.
- Panel D: MK-0941 40 mg Day 13: MK-0941 40 mg before each meal for 13 days. Sampling began after dosing on Day 13. These participants are different from those in Panel C.
- Panel E: MK-0941 60 mg: MK-0941 60 mg before 2 meals each day for 14 days. Sampling began after dosing on Day 13.
Arm/Group | Panel A: MK-0941 10 mg | Panel B: MK-0941 20 mg | Panel C: MK-0941 40 mg Day 7 | Panel D: MK-0941 40 mg Day 13 | Panel E: MK-0941 60 mg
Number analyzed (Participants) | 8 | 7 | 6 | 3 | 4
nM-hr | 2343.29 (253.73) | 3789.25 (1002.05) | 8387.74 (2102.17) | 7673.77 (3616.45) | 8692.07 (2681.37)

3. Secondary Outcome: Maximum Concentration (Cmax) of MK-0941 After Multiple Doses of MK-0941
Time Frame: Up to 72 hours after dosing (up to 24 hours for participants receiving MK0941 60 mg before 2 meals each day)
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Panel A: MK-0941 10 mg | Panel B: MK-0941 20 mg | Panel C: MK-0941 40 mg Day 7 | Panel D: MK-0941 40 mg Day 13 | Panel E: MK-0941 60 mg
Number analyzed (Participants) | 8 | 7 | 6 | 3 | 4
nM | 228.35 (88.54) | 364.96 (151.25) | 841.57 (348.34) | 648.49 (159.73) | 1145.81 (330.56)

4. Secondary Outcome: Time to Maximum Concentration (Tmax) of MK-0941 After Multiple Doses of MK-0941
Time Frame: Up to 72 hours after dosing (up to 24 hours for participants receiving MK0941 60 mg before 2 meals each day)
Measure: Mean (Full Range); unit: hours
Arm/Group | Panel A: MK-0941 10 mg | Panel B: MK-0941 20 mg | Panel C: MK-0941 40 mg Day 7 | Panel D: MK-0941 40 mg Day 13 | Panel E: MK-0941 60 mg
Number analyzed (Participants) | 8 | 7 | 6 | 3 | 4
hours | 1.5 (6.43) [1 to 4] | 1.0 (9.35) [1 to 2] | 1.0 (34.95) [1 to 4] | 1.0 (24.27) [1 to 1] | 2.0 (82.68) [1 to 5]

5. Secondary Outcome: Apparent Terminal Elimination Half-life (T1/2) of MK-0941 After Multiple Doses of MK0941
Time Frame: Up to 72 hours after dosing (up to 24 hours for participants receiving MK0941 60 mg before 2 meals each day)
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Panel A: MK-0941 10 mg Before Each Meal: MK-0941 10 mg before each meal for 5 days. Sampling began after dosing on Day 5.
Arm/Group | Panel A: MK-0941 10 mg Before Each Meal | Panel B: MK-0941 20 mg | Panel C: MK-0941 40 mg Day 7 | Panel D: MK-0941 40 mg Day 13 | Panel E: MK-0941 60 mg
Number analyzed (Participants) | 8 | 7 | 6 | 3 | 4
hours | 10.4 (5.2) | 11.4 (2.2) | 8.4 (6.3) | 10.1 (3.5) | 11.4 (2.1)

6. Secondary Outcome: Concentration of MK-0941 at 24 Hours (C24hr) After Multiple Doses of MK-0941
Time Frame: Up to 72 hours after dosing (up to 24 hours for participants receiving MK0941 60 mg before 2 meals each day)
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Panel A: MK-0941 10 mg | Panel B: MK-0941 20 mg | Panel C: MK-0941 40 mg Day 7 | Panel D: MK-0941 40 mg Day 13 | Panel E: MK-0941 60 mg
Number analyzed (Participants) | 8 | 7 | 6 | 3 | 4
nM | 26.75 (6.43) | 42.99 (9.35) | 95.07 (34.95) | 76.89 (24.27) | 149.30 (82.68)

7. Primary Outcome: Participants Discontinued Because of Any Clinical Adverse Experience
Time Frame: Approximately 30 days after last dose of study drug (14 days for participants receiving MK0941 40 mg before each meal)
Measure: Number; unit: participants
Arm/Group | MK-0941 | Placebo
Number analyzed (Participants) | 52 | 18
participants
  Hyperglycemia | 1 | 0
  All other adverse experiences | 0 | 0

ADVERSE EVENTS:
Time Frame: Approximately 30 days after last dose of study drug (14 days for participants receiving MK-0941 40 mg before each meal)
Arm/Group | MK-0941 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/18
Other Adverse Events (participants affected / at risk) | 27/52 | 11/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MK-0941 (N=52) | Placebo (N=18)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Eye pain (Eye disorders) | 0 | 1
Eye pruritus (Eye disorders) | 1 | 1
Lacrimation increased (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 10 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Dizziness (Nervous system disorders) | 5 | 1
Headache (Nervous system disorders) | 11 | 5
Dysuria (Renal and urinary disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Peripheral coldness (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.